CLINICAL TRIAL: NCT06810375
Title: Erector Spinae Versus Intercostal Nerve Blocks With Liposomal Bupivacaine for Analgesia in Thoracic Surgery
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: George Washington University (Other)
Responsible Party: Principal Investigator, Akhil Patel, MD, Principal Investigator, George Washington University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCR246143
Record Dates: First submitted 2025-01-24; First posted 2025-02-05 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-02

CONDITIONS: Lung Cancers
MeSH Terms: conditions — Lung Neoplasms | interventions — Parapsychology; Dental Occlusion; Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Preoperative Erector Spinae Block (ESB)(Bupivacaine)(Marcaine®) (Active Comparator)
  Interventions: Drug: Erector Spinae (ESP) Block with Bupivacaine (Marcaine®); Drug: Intercostal nerve block
- Intraoperative Intercostal Nerve Block (INB)(Liposomal Bupivacaine)(Exparel®) (Active Comparator)
  Interventions: Drug: Erector Spinae (ESP) Block with Bupivacaine (Marcaine®); Drug: Intercostal nerve block

INTERVENTIONS:
Drug: Erector Spinae (ESP) Block with Bupivacaine (Marcaine®) — preoperative erector spinae block with bupivacaine (Marcaine®)
Drug: Intercostal nerve block — intraoperative intercostal nerve block with liposomal bupivacaine (Exparel®)

SUMMARY:
This clinical trial compares efficacy in postoperative pain management in thoracic surgery between erector spinae block versus liposomal bupivacaine injections.

ELIGIBILITY:
Inclusion Criteria:

* Video assisted pulmonary resection, pleurodesis or decortication

Exclusion Criteria:

* Allergy to local anesthetics
* Patient undergoing bilateral surgery
* Surgery is emergent as deemed by the principal investigator

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2028-02-28 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain control assessment | Up to 48 hours postoperatively
  Study team will assess postoperative pain scores at 6, 12, 24 and 48 hours (Minimum numerical pain score of 0 and a maximum of 10)
Morphine equivalent assessment | Up to 72 hours postoperatively
  Study team will collect information on all administered pain medications to calculate morphine equivalents

SECONDARY OUTCOMES:
Postoperative pain control assessment | Up to 72 hours postoperatively
  Study team will assess postoperative pain scores at 72 hours (Minimum numerical pain score of 0 and a maximum of 10)

CONTACTS AND LOCATIONS:
Locations (1):
- The George Washington University Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No